CLINICAL TRIAL: NCT01443663
Title: Immunogenicity and Safety Study of a 45 Micrograms Dose of Inactivated, Unadjuvanted H5N1 Influenza Vaccine in Prior Recipients of Live Attenuated H5N1 and H7N3 Influenza Vaccines and in H5 and Live Attenuated Vaccine Naïve Individuals
Brief Title: Evaluating the Safety and Immune Response to an H5N1 Influenza Vaccine in People Who Have Previously Received an H5N1 or H7N3 Influenza Vaccine and in People Who Have Never Received a Live Attenuated Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIR 277
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: H5N1 Influenza

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Previously Received H5N1 VN 04 ca Vaccine) (Experimental): Participants will have previously received two doses of 10^7.5 tissue culture infectious dose (TCID)50 of H5N1 A/VN/1203/04 x A/AA/6/60 ca LAIV (H5N1 VN 04 ca). In this study, they will receive one dose of the H5N1 vaccine at baseline.
  Interventions: Biological: H5N1 Vaccine
- Group 2 (Previously Received H5N1 HK 03 ca Vaccine) (Experimental): Participants will have previously received two doses of 10^7.5 TCID50 of H5N1 A/HK/213/03 x A/AA/6/60 ca LAIV (H5N1 HK 03 ca). In this study, they will receive one dose of the H5N1 vaccine at baseline.
  Interventions: Biological: H5N1 Vaccine
- Group 3 (Previously Received H7N3 ca Vaccine) (Experimental): Participants will have previously received two doses of 10^7.5 TCID50 of H7N3 A/ck/BC/CN-6/04 x A/AA/6/60 ca LAIV (H7N3 ca). In this study, they will receive one dose of the H5N1 vaccine at baseline.
  Interventions: Biological: H5N1 Vaccine
- Group 4 (Have Not Previously Received LAIV) (Experimental): Participants will have not previously received an LAIV of any kind. In this study, they will receive one dose of the H5N1 vaccine at baseline.
  Interventions: Biological: H5N1 Vaccine
- Group 5 (Have Not Previously Received LAIV) (Experimental): Participants will have not previously received an LAIV of any kind. In this study, they will receive two doses of the H5N1 vaccine at baseline and Day 28.
  Interventions: Biological: H5N1 Vaccine

INTERVENTIONS:
Biological: H5N1 Vaccine — Vaccine will be administered intramuscularly (IM) in the deltoid muscle at baseline for participants in Groups 1-4 and at baseline and Day 28 for participants in Group 5.

SUMMARY:
H5N1 is an influenza virus that has the potential to cause an influenza pandemic. This study will evaluate the safety and immune response to an H5N1 influenza vaccine in people who have previously received one of two versions of an H5N1 vaccine or have previously received an H7N3 vaccine and in people who have not previously received any live attenuated influenza vaccine (LAIV).

DETAILED DESCRIPTION:
Avian influenza viruses, including H1N1 and H5N1, are capable of causing an influenza pandemic. The 2009 H1N1 pandemic caused approximately 10,000 deaths in the United States, and H1N1 and H5N1 influenza outbreaks have been observed in countries around the world. Previous studies have shown that people who received an H5N1 vaccine and then received another H5N1 vaccine years later had a greater antibody response than people who only received a single vaccination. This study will evaluate the safety and immune response to an inactivated H5N1 vaccine in healthy adults who have previously received two doses of the H5N1 VN 04 ca vaccine or the H5N1 HK 03 ca vaccine or who have previously received two doses of the H7N3 ca vaccine, which is another avian influenza vaccine. The study will also enroll people who have not previously received any LAIV.

Participants who previously received an H5N1 or H7N3 vaccine will receive one injection of the H5N1 vaccine at baseline. Participants who have not received any previous LAIV will be randomly assigned to receive either one dose or two doses of the H5N1 vaccine. At a baseline study visit, participants will undergo a medical history review, physical examination, blood collection, vital sign measurements, and a pregnancy test for females. All participants will then receive one injection of the vaccine in the upper arm. After receiving the vaccine, participants will remain in the clinic for 30 minutes for observation and monitoring. All participants will attend additional study visits at Days 3 and 7. Participants who are assigned to receive one vaccination will also attend study visits at Days 28, 56, and 180. Participants who are assigned to receive two vaccinations will attend study visits at Days 28 (at which time they will receive the second vaccination), 35, 56, 84, and 208. Select baseline study procedures will occur at the follow-up study visits.

ELIGIBILITY:
Inclusion Criteria:

* In general good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator
* Available for the duration of the trial
* Willing to participate in the study as evidenced by signing the informed consent document
* Willing to allow storage and testing of laboratory samples for future research
* Received two doses of live attenuated H5N1 or H7N3 vaccine in a prior trial (Study Groups 1, 2, and 3) or LAIV and H5 naïve (Study Groups 4 and 5)
* Willing to forego seasonal LAIV for the duration of the trial (until 6 months after the last vaccination)
* Female participants must agree to use effective birth control methods for the duration of the study. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Pregnant, as determined by a positive beta-human choriogonadotropin (HCG) test
* Currently breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the 12 months prior to study entry
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* History of anaphylaxis
* History of life-threatening reaction to prior influenza vaccine
* Current diagnosis of asthma or reactive airway disease (within the 2 years prior to study entry)
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory Western blot tests for HIV-1
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay [RIBA]) for hepatitis C virus (HCV)
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA
* Known immunodeficiency syndrome
* History of Guillain-Barré syndrome
* Use of chronic oral or intravenous administration (greater than or equal to 14 days) of immunosuppressive doses of steroids, i.e., prednisone greater than 10 mg per day, immunosuppressants or other immune-modifying drugs within 30 days of starting this study
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products

In addition to the above, participants in the H5 and LAIV-naïve groups must also not experience any of the following:

* Previous enrollment in an H5 influenza vaccine trial or in any study of an avian influenza (AI) vaccine
* Seropositive to the H5N1 influenza A virus (serum HI titer greater than 1:8)
* Previous receipt of FluMist or any intranasal live attenuated influenza vaccine

Ages: 22 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Characterize the kinetics and magnitude of the antibody response (measured by hemagglutination inhibition assay [HI] and microneutralization assay [MN]) to a single 45 micrograms dose of H5N1 vaccine | Measured through the 6 months following participants' last vaccination

SECONDARY OUTCOMES:
Assess the reactogenicity of the H5N1 vaccine in previous recipients of LAIV | Measured through the 6 months following participants' last vaccination
  Reactogenicity will be followed for 7 days; serious adverse events (SAEs) will be followed for 6 months after the last immunization.
Assess the immune response to the inactivated H5N1 vaccine (A/VN/1203/04) | Measured through the 6 months following participants' last vaccination
  Immune response will be assessed via the following:
  1. Evaluation of memory B-cell responses to H5N1 by enzyme-linked immunosorbent spot (ELISPOT)
  2. Evaluation of HI antibody responses to heterologous non-Clade 1 H5N1 viruses
  3. Evaluation of T-cell mediated responses to H5N1 influenza viruses to the following:
     1. Clade 1 H5N1 viruses
     2. Heterologous cross-clade H5N1 viruses

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R. Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Centers for Immunization Research (CIR) - John Hopkins Bloomburg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Goji NA, Nolan C, Hill H, Wolff M, Noah DL, Williams TB, Rowe T, Treanor JJ. Immune responses of healthy subjects to a single dose of intramuscular inactivated influenza A/Vietnam/1203/2004 (H5N1) vaccine after priming with an antigenic variant. J Infect Dis. 2008 Sep 1;198(5):635-41. doi: 10.1086/590916. PMID 18694338
- [Background] Galli G, Hancock K, Hoschler K, DeVos J, Praus M, Bardelli M, Malzone C, Castellino F, Gentile C, McNally T, Del Giudice G, Banzhoff A, Brauer V, Montomoli E, Zambon M, Katz J, Nicholson K, Stephenson I. Fast rise of broadly cross-reactive antibodies after boosting long-lived human memory B cells primed by an MF59 adjuvanted prepandemic vaccine. Proc Natl Acad Sci U S A. 2009 May 12;106(19):7962-7. doi: 10.1073/pnas.0903181106. Epub 2009 Apr 27. PMID 19416838
- [Derived] Talaat KR, Luke CJ, Khurana S, Manischewitz J, King LR, McMahon BA, Karron RA, Lewis KD, Qin J, Follmann DA, Golding H, Neuzil KM, Subbarao K. A live attenuated influenza A(H5N1) vaccine induces long-term immunity in the absence of a primary antibody response. J Infect Dis. 2014 Jun 15;209(12):1860-9. doi: 10.1093/infdis/jiu123. Epub 2014 Mar 5. PMID 24604819